## Effectiveness of hypnoanalgesia for dermatological surgery in children: Randomised clinical trial

## NCT CHT00028

Document Date: March 15, 2019

Statistical plan

For the descriptive analysis, central tendency and dispersion measures will be used (median and 25<sup>th</sup> to 75<sup>th</sup> percentiles, P<sub>25-75</sub>) for quantitative variables, and absolute and relative frequencies for qualitative ones.

The comparison of the outcome measures between the intervention group and the control group will be carried out by means of non-parametric tests: chi-square and Fisher's exact test for qualitative outcome measures, and Mann-Whitney's U for the quantitative ones.

An age-based subgroup analysis will be conducted (under 7 years and over).

The significance level will be set at a value of p<0.05 and the analysis will be carried out with Excel®.

A sample of 30 patients was calculated to detect a 40 mg dose difference between the two groups, with a risk  $\alpha$  of 0.05 and a risk  $\beta$  of 0.20 in a bilateral contrast and assuming a common standard deviation of 33.3 and a loss to follow-up rate of 10%.